CLINICAL TRIAL: NCT06092944
Title: Clinical Study of Rhomboid Intercostal and Subserratum Plane Block for Postoperative Analgesia in Minimally Invasive Esophagectomy
Brief Title: Rhomboid Intercostal and Subserratum Plane Block for Minimally Invasive Esophagectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luo Fuchao (Other)
Responsible Party: Sponsor-Investigator, Luo Fuchao, principal, Fuling Central Hospital of Chongqing City
Organization: Fuling Central Hospital of Chongqing City (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RISS
Record Dates: First submitted 2023-09-27; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Esophagus Cancer
Keywords: Rhomboid intercostal and subserratum plane block; Ultrasound-guided; Postoperative analgesia; Minimally invasive esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Catheterization; Nerve Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- continuous RISS group (Experimental): Patients were given continuous RISS plane block in addition to patient controlled intravenous analgesia.
  Interventions: Procedure: Catheterization; Procedure: Single nerve block; Procedure: Continuous nerve block; Procedure: PCIA
- single RISS group (Experimental): Patients were given single RISS plane block in addition to patient controlled intravenous analgesia.
  Interventions: Procedure: Single nerve block; Procedure: PCIA
- PCIA group (Active Comparator): Patients were given patient controlled intravenous analgesia.
  Interventions: Procedure: PCIA

INTERVENTIONS:
Procedure: Catheterization — Before the operation,the patient was placed in the left lateral position.The catheter（soft tip epidural catheter 20-gauge-100 cm） was placed at the rhomboid-intercostal plane under ultrasound guidance at the T5-T6 level, followed by ultrasound-guided catheter placed in the anterior serrated muscle plane at the T7-9 level。
  Arms: continuous RISS group
Procedure: Single nerve block — Before the operation,40milliliters of 0.3% ropivacaine was injected into the rhomboid-intercostal fascia plane and anterior serrated muscle plane respectively under the guidance of ultrasound.
  Arms: continuous RISS group; single RISS group
Procedure: Continuous nerve block — After surgery,local anesthetics were injected continuously through catheters.Local anesthetic formula:Ropivacaine 300mg + normal saline, prepared into 150milliliters liquid, background dose 2milliliters/h.
  Arms: continuous RISS group
Procedure: PCIA — After surgery, the patient was given controlled intravenous analgesia. Analgesic pump drug formula:Sufentanil 50ug+ Dezocine 20mg+ Granisetron 10mg+150milliliters saline, continuous dose of 2milliliters/h intravenous pump, single injection dose of 2milliliters, locking time of 20 min

SUMMARY:
The objective is to investigate the safety and effectiveness of rhomboid intercostal and subserratum plane (RISS) block for postoperative analgesia after minimally invasive McKeown esophagectomy (MIE-McKeown).

DETAILED DESCRIPTION:
Rhomboid intercostal and subserratum plane block (RISS) is a nerve block technique in which local anesthetics are injected into the rhomboid-intercostal muscle planes and the serratus anterius-intercostal muscle planes, and the intercostal nerve is blocked by diffusion of local anesthetics. It is confirmed that RISS can provide analgesia not only in the front half of the chest, but also in the upper abdomen. However, the efficacy of RISS in minimally invasive surgery for esophageal cancer has not been proven. The investigators placed catheters on the RISS plane and continuously injected local anesthetics to investigate whether RISS is effective and safe in minimally invasive esophageal cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients received MIE-McKeown surgery and were confirmed by postoperative pathology; Age 18-75 years old
* body mass index (BMI) : 18.5~23.9kg/m2;
* American Society of Anesthesiologists (ASA) grade: Ⅰ~Ⅱ;
* Clear consciousness, no cognitive impairment;
* Patients informed to participate in the study and signed informed consent.

Exclusion Criteria:

* Infection of the puncture site, abnormal platelet or coagulation function;
* Patients with drug allergy involved in this study;
* Long-term use of analgesic, sedative drugs or a history of heavy drinking;
* Patients with chronic painful diseases;
* With severe heart, liver, kidney and lung dysfunction;
* Infectious diseases, blood, immune, circulatory system diseases; -Communication barriers, can not cooperate with the scale assessment; -
* Other situations not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Analgesic effect | 2, 6, 12, 24, and 48 hours after surgery
  patient will be asked to rate their pain level at rest and cough respectively using visual analogue scale（VAS）.(0 being no pain, 10 being worst pain imaginable)
mean arterial pressure (MAP) | before anesthesia induction (T0)， before skin incision（T1）， 5 minutes after skin incision
  The mean arterial pressure (MAP)on the monitor at different times was recorded.
Heart rate (HR) | before anesthesia induction (T0)， before skin incision（T1）， 5 minutes after skin incision
  The Heart rate (HR)on the monitor at different times was recorded.

SECONDARY OUTCOMES:
dizziness | 24hours after surgery
  The occurrence of dizziness was recorded
lethargy | 24hours after surgery
  The occurrence of lethargy was recorded
nausea or vomiting | 24hours after surgery
  The occurrence of nausea /vomiting was recorded
hypotension | 24hours after surgery
  The occurrence of hypotension was recorded
respiratory depression | 24hours after surgery
  The occurrence of respiratory depression was recorded
urinary retention | 24hours after surgery
  The occurrence of urinary retention was recorded
Analgesia satisfaction | 24hours after surgery
  patient will be asked to rate their Satisfaction with analgesia using verbal rating scales (VRS) .Scores from 1 to 5 represent very dissatisfied, not satisfied, basically satisfied, relatively satisfied, and very satisfied with the analgesic effect, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Luo fuchao, MD, Principal Investigator — Chongqing University Fuling Hospital
Locations (1):
- FulingCH, Chongqing, China

IPD SHARING:
Plan to Share IPD: No